CLINICAL TRIAL: NCT05293795
Title: The Impact of 3D Ultrasound on Maternal-Fetal Attachment Among African American Women
Brief Title: 3D U/S Maternal Fetal Bonding in African American Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2002129
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Maternal-Fetal Relations; Maternal Behavior

STUDY DESIGN:
Intervention Model Description: 3D ultrasound and picture of ultrasound or 3D ultrasound and printed model of fetal face and normal controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3d printed model (Active Comparator): Mother r is given 3D printed model of fetus' face
  Interventions: Behavioral: 3D printed model
- Placebo (Placebo Comparator): Mother is given printed picture of 3D ultrasound of fetus
  Interventions: Behavioral: Placebo
- Control (No Intervention): Standard of Care

INTERVENTIONS:
Behavioral: 3D printed model — Mother is given 3D printed model of fetus' face
  Arms: 3d printed model
Behavioral: Placebo — Mother is given a picture of 3D ultrasound of fetus
  Arms: Placebo

SUMMARY:
To determine whether 3D models of fetus' face created from 3D ultrasound will increase maternal and paternal attachment, lower stress, anxiety and depression and have improved life-style choices during pregnancy in African-American women.One-third of participants will receive 3D model and complete questionnaires, one-third will receive a picture of 3D ultrasound of their baby and complete questionnaires, and one-third will only complete the questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Age - Female 19-45 years of age
* Fluent in English
* African American
* Currently pregnant (between 26- and 31-weeks' gestation)
* Have normal 20-week ultrasound

Exclusion Criteria:

* Having received more than 3 ultrasounds prior to study
* Medical need for additional ultrasounds
* Multiple fetuses
* > 31 weeks gestation
* Is not African American
* Is not fluent in English

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female gender assigned at birth only
Enrollment: 144 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Maternal Antenatal Attachment Scale (MAAS) | 5 minutes
  The MAAS is a 19 item questionnaire measuring maternal-fetal attachment. Each item has five answer choices scored from 1 low attachment to 5 high attachment such that the total score ranges from 19 to 95. The measure also includes two subscales: (1) Quality of Attachment has 10 items with a range of 10-50 and measures the quality of the mother's attachment to her fetus.
  (2) Time measures the time spent in attachment mode (or intensity of preoccupation) and consists of 8 items for a range of 8 to 40. (for clarity one item included in the total score is not included in either subscale.)
Maternal Anxiety | 3 minutes
  7-question Generalized Anxiety Disorder questionnaire (GAD-7) will be administered
Maternal Depression | 3 minutes
  9-question Patient Health Questionnaire (PHQ-9) will be administered
Maternal Stress | 3 minutes
  11-question Pregnancy-Related Anxiety Questionnaire-Revised (PRAQ-R2) will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Kalata, MD, MPH, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No